CLINICAL TRIAL: NCT03984838
Title: A Phase I, Open-label, Single-dose Study to Investigate the Pharmacokinetics, Safety and Tolerability of Dolutegravir + Rilpivirine (JULUCA™) 50 mg/25 mg Tablets in Healthy Participants of Japanese Descent
Brief Title: Study to Evaluate Pharmacokinetics, Safety and Tolerability of Dolutegravir and Rilpivirine (JULUCA™) 50 Milligram (mg)/25 mg Tablets in Healthy Subjects of Japanese Descent
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 212312
Record Dates: First submitted 2019-06-10; First posted 2019-06-13 (Actual); Results first posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-06

CONDITIONS: HIV Infections
Keywords: Dolutegravir, Rilpivirine, HIV infection, Fixed-dose combination, Japanese, Pharmacokinetics
MeSH Terms: conditions — HIV Infections | interventions — dolutegravir, rilpivirine drug combination; dolutegravir; Rilpivirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Subjects receiving Dolutegravir and Rilpivirine FDC (Experimental): Subjects will receive Dolutegravir/Rilpivirine 50mg/25mg fixed dose combination (FDC) tablet as a single oral dose in a fed state.
  Interventions: Drug: JULUCA (Dolutegravir and Rilpivirine) 50mg/25mg FDC tablet

INTERVENTIONS:
Drug: JULUCA (Dolutegravir and Rilpivirine) 50mg/25mg FDC tablet — JULUCA tablets will be administered orally once daily with a meal. It will be available as a fixed dose combination of Dolutegravir 50mg and Rilpivirine 25mg.

SUMMARY:
Dolutegravir (DTG), a human immunodeficiency virus (HIV)-1 integrase inhibitor (INI), and Rilpivirine (RPV), a non-nucleoside HIV-1 reverse transcriptase inhibitor (NNRTI), are each approved in the United States (US), European Union, and other countries for the treatment of HIV-1 infection. JULUCA is a combination of Dolutegravir and Rilpivirine indicated for the treatment of HIV-1 infection in antiretroviral (ARV) experienced adult subjects who are switching from their current antiretroviral treatment to the 2-drug combination. Although, the pharmacokinetics (PK), safety and tolerability of DTG/RPV (50 milligram [mg]/25mg) fixed-dose combination (FDC) tablets have been extensively studied, these parameters have not been assessed exclusively in Japanese subjects. This study will evaluate the pharmacokinetics, safety and tolerability of a single dose DTG/RPV 50 mg/25 mg FDC in a healthy adult Japanese population to support a post-approval commitment for DTG/RPV 50 mg/25 mg FDC in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 to 55 years of age, at the time of signing the informed consent
* Subjects who were born in Japan with 4 ethnic Japanese grandparents. Subjects who have not lived outside Japan for more than 10 years and who are Japanese passport holders (current or expired)
* Subjects who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring (history and electrocardiogram [ECG])
* Subjects with body weight >=50 kilogram (kg) (110 pounds) for men and >=45kg (99 pounds) for women and body mass index (BMI) within the range 18.5-31.0 kg per square meter (kg/m^2)
* Male or female subjects; Male subjects with no specific restrictions
* A female subject is eligible to participate if she is not pregnant or breastfeeding, and not a woman of childbearing potential (WOCBP)
* The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy
* Subjects capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol

Exclusion Criteria:

* Subjects with history of current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention or interfering with the interpretation of data
* Subjects with abnormal blood pressure (as determined by the investigator)
* Subjects with alanine transaminase (ALT) >1.5 times upper limit of normal (ULN)
* Subjects with bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* Subjects with current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Subjects with QTcF >460 millisecond (msec)(Based on the average of the 12-Lead-electrocardiogram (ECG) triplicate readings obtained at Screening) (Note: The QTc is the QT interval corrected for heart rate according to Fridericia's formula (QTcF), and/or another method, machine-read or manually over-read. The specific formula that will be used to determine eligibility and discontinuation for an individual subject should be determined prior to initiation of the study. In other words, several different formulae cannot be used to calculate the QTc for an individual subject and then the lowest QTc value used to include or discontinue the subject from the trial)
* Subjects with past or intended use of over-the-counter or prescription medication including herbal medications within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to dosing. Acetaminophen, at doses of <=2 grams per day, is allowed for use any time during the study
* Participation in the study would result in loss of blood or blood products in excess of 500 milliliter (mL) within 56 days
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day
* Current enrollment or past participation within the last 30 days before signing of consent in any other clinical study involving an investigational study intervention or any other type of medical research
* Subjects with presence of Hepatitis B surface antigen (HBsAg) at screening or within 3 months prior to first dose of study intervention
* Subjects with positive Hepatitis C antibody test result at screening or within 3 months prior to first dose of study intervention (Note: Subjects with positive Hepatitis C antibody due to prior resolved disease can be enrolled, only if a confirmatory negative Hepatitis C RNA test is obtained)
* Subjects with positive Hepatitis C RNA test result at screening or within 3 months prior to first dose of study intervention (Note: Test is optional and subjects with negative Hepatitis C antibody test are not required to also undergo Hepatitis C RNA testing)
* Subjects with positive pre-study drug or alcohol screen
* Subjects with positive human immunodeficiency virus (HIV) antibody test
* Subjects with regular use of known drugs of abuse
* Subjects with creatinine clearance (CrCL) <60 milliliter per minute
* Employment with Janssen, ViiV, GlaxoSmithKline(GSK), or with the Investigator or study site, with direct involvement in the proposed study or other studies under the direction of that Investigator or study site, as well as family members of the employees or the Investigator
* Subjects with urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products (e.g. nicotine patches or vaporizing devices) within 6 months prior to screening
* Subjects with regular alcohol consumption within 6 months prior to the study defined as: An average weekly intake of >14 units for males or >7 units for females. One unit is equivalent to 8 gram of alcohol: a half-pint (approximately 240mL) of beer, 1 glass (125mL) of wine or 1 (25mL) measure of spirits
* Subjects with sensitivity to heparin or heparin-induced thrombocytopenia
* Subjects with sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2019-08-13 (Actual); Study Completion 2019-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The was a single dose, open-label study in healthy Japanese participants for the evaluation of pharmacokinetics (PK), safety and tolerability of fixed dose combination (FDC) tablet of Dolutegravir (DTG)/Rilpivirine (RPV) 50 milligrams (mg)/ 25 mg
Pre-assignment Details: A total of 16 participants were enrolled in the study
Groups:
- DTG/RPV 50mg/25mg FDC: Healthy participants were administered single oral FDC tablet of DTG/RPV 50mg/25mg on Day 1 in fed state
Period: Overall Study
Arm/Group | DTG/RPV 50mg/25mg FDC
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.6 (9.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese Heritage/East Asian | 16

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration (AUC) Time Curve From Time Zero Extrapolated to Infinite Time (AUC [0-infinity]) of DTG
Description: Blood samples were collected at indicated time-points for analysis of AUC (0-infinity) of DTG. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, 24, 48, 72, and 120 hours post-dose
Population: PK Population included all participants in the Safety Population (participants who were enrolled in the study and received at least one dose of study drug) for whom a PK sample was obtained and had evaluable PK assay results.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Hours*micrograms per milliliter | 90.9402 (26.2)

2. Primary Outcome: AUC (0-infinity) of RPV
Description: Blood samples were collected at indicated time-points for analysis of AUC (0-infinity) of RPV. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, 24, 48, 72, 120, 168, 216, and 264 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Hours*nanogram per milliliter | 4027.9415 (29.0)

3. Primary Outcome: Area Under the Concentration Time Curve From Time Zero to Last Time of Quantifiable Concentration (AUC [0-t]) of DTG
Description: Blood samples were collected at indicated time-points for analysis of AUC (0-t) of DTG. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, 24, 48, 72, and 120 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Hours*micrograms per milliliter | 89.1993 (26.8)

4. Primary Outcome: AUC (0-t) of RPV
Description: Blood samples were collected at indicated time-points for analysis of AUC (0-t) of RPV. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, 24, 48, 72, 120, 168, 216, and 264 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Hours*nanogram per milliliter | 3920.9404 (29.1)

5. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of DTG
Description: Blood samples were collected at indicated time-points for analysis of Cmax of DTG. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, 24, 48, 72, and 120 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Nanograms per milliliter | 4108.5 (15.0)

6. Primary Outcome: Cmax of RPV
Description: Blood samples were collected at indicated time-points for analysis of Cmax of RPV. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, 24, 48, 72, 120, 168, 216, and 264 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Nanogram per milliliter | 136.10 (34.3)

7. Primary Outcome: Absorption Lag Time (Tlag) of DTG
Description: Blood samples were collected at indicated time-points for analysis of tlag of DTG. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, 24, 48, 72, and 120 hours post-dose
Population: PK Population
Measure: Median (Full Range); unit: Hours
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Hours | 0.0 [0 to 1]

8. Primary Outcome: Tlag of RPV
Description: Blood samples were collected at indicated time-points for analysis of tlag of RPV. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, 24, 48, 72, 120, 168, 216, and 264 hours post-dose
Population: PK Population
Measure: Median (Full Range); unit: Hours
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Hours | 0.5 [0 to 2]

9. Primary Outcome: Time to Reach Maximum Observed Concentration (Tmax) of DTG
Description: Blood samples were collected at indicated time-points for analysis of tmax of DTG. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, 24, 48, 72, and 120 hours post-dose
Population: PK Population
Measure: Median (Full Range); unit: Hours
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Hours | 3.0085 [1.002 to 5.003]

10. Primary Outcome: Tmax of RPV
Description: Blood samples were collected at indicated time-points for analysis of tmax of RPV. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, 24, 48, 72, 120, 168, 216, and 264 hours post-dose
Population: PK Population
Measure: Median (Full Range); unit: Hours
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Hours | 4.4976 [3.503 to 5.999]

11. Primary Outcome: Time of Last Quantifiable Concentration (Tlast) of DTG
Description: Blood samples were collected at indicated time-points for analysis of tlast of DTG. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, 24, 48, 72, and 120 hours post-dose
Population: PK Population
Measure: Median (Full Range); unit: Hours
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Hours | 120.0854 [71.818 to 145.015]

12. Primary Outcome: Tlast of RPV
Description: Blood samples were collected at indicated time-points for analysis of tlast of RPV. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, 24, 48, 72, 120, 168, 216, and 264 hours post-dose
Population: PK Population
Measure: Median (Full Range); unit: Hours
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Hours | 214.5819 [120.570 to 265.502]

13. Primary Outcome: Elimination Half-life (t1/2) of DTG
Description: Blood samples were collected at indicated time-points for analysis of t1/2 of DTG. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, 24, 48, 72, and 120 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Hours | 17.3135 (15.6)

14. Primary Outcome: T1/2 of RPV
Description: Blood samples were collected at indicated time-points for analysis of t1/2 of RPV. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, 24, 48, 72, 120, 168, 216, and 264 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Hours | 37.2571 (33.7)

15. Primary Outcome: Apparent Elimination Rate Constant (Lambda z) of DTG
Description: Blood samples were collected at indicated time-points for analysis of lambda z of DTG. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, 24, 48, 72, and 120 hours post-dose
Population: PK Population
Measure: Mean (Standard Deviation); unit: Per hour
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Per hour | 0.0405 (0.00604)

16. Primary Outcome: Lambda z of RPV
Description: Blood samples were collected at indicated time-points for analysis of lambda z of RPV. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, 24, 48, 72, 120, 168, 216, and 264 hours post-dose
Population: PK Population
Measure: Mean (Standard Deviation); unit: Per hour
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Per hour | 0.0196 (0.00674)

17. Primary Outcome: Percentage of AUC(0-infinity) That Was Extrapolated (%AUCex) of DTG
Description: Blood samples were collected at indicated time-points for analysis of percentage AUCex of DTG. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, 24, 48, 72, and 120 hours post-dose
Population: PK Population
Measure: Mean (Standard Deviation); unit: Percentage of AUCex
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Percentage of AUCex | 1.9065 (1.28407)

18. Primary Outcome: Percentage AUCex of RPV
Description: Blood samples were collected at indicated time-points for analysis of percentage AUCex of RPV. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, 24, 48, 72, 120, 168, 216, and 264 hours post-dose
Population: PK Population
Measure: Mean (Standard Deviation); unit: Percentage of AUCex
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Percentage of AUCex | 2.6501 (1.14962)

19. Primary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero to 24 Hours (AUC[0-24]) of DTG
Description: Blood samples were collected at indicated time-points for analysis of AUC(0-24) of DTG. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, and 24 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Hours*micrograms per milliliter | 54.9466 (20.4)

20. Primary Outcome: AUC (0-24) of RPV
Description: Blood samples were collected at indicated time-points for analysis of AUC (0-24) of RPV. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, and 24 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Hours*nanograms per milliliter | 1420.2525 (24.8)

21. Primary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero to 72 Hours (AUC[0-72]) of DTG
Description: Blood samples were collected at indicated time-points for analysis of AUC(0-72) of DTG. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, 24, 48, and 72 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Hours*micrograms per milliliter | 85.3534 (24.3)

22. Primary Outcome: AUC (0-72) of RPV
Description: Blood samples were collected at indicated time-points for analysis of AUC (0-72) of RPV. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Hours*nanograms per milliliter | 2886.6035 (22.7)

23. Primary Outcome: Apparent Oral Clearance (CL/F) of DTG
Description: Blood samples were collected at indicated time-points for analysis of CL/F of DTG. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, 24, 48, 72, and 120 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Liters per hour | 0.5498 (26.2)

24. Primary Outcome: CL/F of RPV
Description: Blood samples were collected at indicated time-points for analysis of CL/F of RPV. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, 24, 48, 72, 120, 168, 216, 264 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Liters per hour | 6.2066 (29.0)

25. Primary Outcome: Apparent Oral Volume of Distribution (Vz/F) of DTG
Description: Blood samples were collected at indicated time-points for analysis of Vz/F of DTG. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, 24, 48, 72, and 120 hours post-dose
Population: PK Population
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Liters | 14.0079 (2.81380)

26. Primary Outcome: Vz/F of RPV
Description: Blood samples were collected at indicated time-points for analysis of Vz/F of RPV. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, 24, 48, 72, 120, 168, 216, and 264 hours post-dose
Population: PK Population
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Liters | 347.3276 (99.96058)

27. Primary Outcome: Last Quantifiable Concentration (Ct) of DTG
Description: Blood samples were collected at indicated time-points for analysis of Ct of DTG. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, 24, 48, 72, and 120 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Nanograms per milliliter | 54.59 (82.1)

28. Primary Outcome: Ct of RPV
Description: Blood samples were collected at indicated time-points for analysis of Ct of RPV. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, 24, 48, 72, 120, 168, 216, and 264 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Nanograms per milliliter | 1.836 (30.4)

29. Primary Outcome: Concentration at 24-hour Post-dose (C24) of DTG
Description: Blood samples were collected at indicated time-points for analysis of C24 of DTG. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: At 24 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Nanograms per milliliter | 1453.6 (25.6)

30. Primary Outcome: C24 of RPV
Description: Blood samples were collected at indicated time-points for analysis of C24 of RPV. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: At 24 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Nanograms per milliliter | 43.35 (22.1)

31. Secondary Outcome: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. A SAE is defined as any untoward medical occurrence that, at any dose: results in death and is life-threatening; which requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent disability or incapacity and birth defect or congenital anomaly, or any other situation that require medical or scientific judgment.
Time Frame: Up to Day 18
Population: Safety Population included participants who were enrolled in the study and received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Participants
  AE | 2
  SAE | 0

32. Secondary Outcome: Change From Baseline in Neutrophil, Lymphocyte, Leukocyte, Monocyte, Eosinophil, Basophil and Platelet Count
Description: Blood samples were collected at indicated time-points for analysis of hematology parameters like platelet count, neutrophils, lymphocytes, leukocyte, monocytes, eosinophils and basophils. Baseline was defined as Day -1. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1) and Day 3
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Giga cells per liter
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Giga cells per liter
  Basophils | -0.03 (0.045)
  Eosinophils | -0.04 (0.089)
  Leukocytes | -0.16 (1.016)
  Lymphocytes | -0.03 (0.445)
  Monocytes | -0.04 (0.081)
  Platelets | 5.4 (18.85)
  Neutrophils | -0.06 (0.788)

33. Secondary Outcome: Absolute Values of Neutrophil, Lymphocyte, Leukocyte, Monocyte, Eosinophil, Basophil and Platelet Count
Description: Blood samples were collected at indicated time-points for analysis of hematology parameters like platelet count, neutrophils, lymphocytes, monocytes, leukocyte, eosinophils and basophils. Baseline was defined as Day -1.
Time Frame: Baseline (Day -1) and Day 3
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Giga cells per liter
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Giga cells per liter
  Basophils, Baseline (Day -1) | 0.04 (0.050)
  Basophils, Day 3 | 0.01 (0.034)
  Eosinophils, Baseline (Day -1) | 0.20 (0.110)
  Eosinophils, Day 3 | 0.16 (0.063)
  Leukocytes, Baseline (Day -1) | 5.76 (1.238)
  Leukocytes, Day 3 | 5.59 (1.433)
  Lymphocytes, Baseline (Day -1) | 1.84 (0.407)
  Lymphocytes, Day 3 | 1.82 (0.565)
  Monocytes, Baseline (Day -1) | 0.45 (0.126)
  Monocytes, Day 3 | 0.41 (0.141)
  Platelets, Baseline (Day -1) | 233.3 (43.24)
  Platelets, Day 3 | 238.6 (47.88)
  Neutrophils, Baseline (Day -1) | 3.21 (0.973)
  Neutrophils, Day 3 | 3.16 (1.001)

34. Secondary Outcome: Change From Baseline in Hemoglobin Level
Description: Blood samples were collected at indicated timepoints for analysis of hematology parameter like hemoglobin. Baseline was defined as Day -1. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1) and Day 3
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Grams per liter | 10.1 (7.33)

35. Secondary Outcome: Absolute Values of Hemoglobin Level
Description: Blood samples were collected at indicated timepoints for analysis of hematology parameter like hemoglobin. Baseline was defined as Day -1.
Time Frame: Baseline (Day -1) and Day 3
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Grams per liter
  Baseline (Day -1) | 140.9 (15.92)
  Day 3 | 151.0 (15.19)

36. Secondary Outcome: Change From Baseline in Hematocrit Level
Description: Blood samples were collected at indicated timepoints for analysis of hematology parameter like hematocrit. Baseline was defined as Day -1. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1) and Day 3
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Proportion of red blood cells in blood | 0.0308 (0.01967)

37. Secondary Outcome: Absolute Values of Hematocrit Level
Description: Blood samples were collected at indicated timepoints for analysis of hematology parameter like hematocrit. Baseline was defined as Day -1.
Time Frame: Baseline (Day -1) and Day 3
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Proportion of red blood cells in blood
  Baseline (Day -1) | 0.4248 (0.04060)
  Day 3 | 0.4556 (0.04087)

38. Secondary Outcome: Change From Baseline in Erythrocytes
Description: Blood samples were collected at indicated timepoints for analysis of hematology parameter like erythrocytes. Baseline was defined as Day -1. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1) and Day 3
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Trillion cells per liter | 0.358 (0.2112)

39. Secondary Outcome: Absolute Values of Erythrocytes
Description: Blood samples were collected at indicated timepoints for analysis of hematology parameter like erythrocytes. Baseline was defined as Day -1.
Time Frame: Baseline (Day -1) and Day 3
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Trillion cells per liter
  Baseline (Day -1) | 4.688 (0.5299)
  Day 3 | 5.046 (0.4994)

40. Secondary Outcome: Change From Baseline in Mean Corpuscular Hemoglobin (MCH)
Description: Blood samples were collected at indicated timepoints for analysis of hematology parameter like MCH. Baseline was defined as Day -1. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1) and Day 3
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Picograms | -0.10 (0.303)

41. Secondary Outcome: Absolute Values of MCH
Description: Blood samples were collected at indicated timepoints for analysis of hematology parameter like MCH. Baseline was defined as Day -1.
Time Frame: Baseline (Day -1) and Day 3
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Picograms
  Baseline (Day -1) | 30.04 (1.288)
  Day 3 | 29.94 (1.275)

42. Secondary Outcome: Change From Baseline in Mean Corpuscular Volume (MCV)
Description: Blood samples were collected at indicated timepoints for analysis of hematology parameter like MCV. Baseline was defined as Day -1. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1) and Day 3
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Femtoliters | -0.43 (0.849)

43. Secondary Outcome: Absolute Values of MCV
Description: Blood samples were collected at indicated timepoints for analysis of hematology parameter like MCV. Baseline was defined as Day -1.
Time Frame: Baseline (Day -1) and Day 3
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Femtoliters
  Baseline (Day -1) | 90.87 (3.593)
  Day 3 | 90.44 (3.522)

44. Secondary Outcome: Change From Baseline in Reticulocytes
Description: Blood samples were collected at indicated timepoints for analysis of hematology parameter like reticulocytes. Baseline was defined as Day -1. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1) and Day 3
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Percentage of reticulocytes
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Percentage of reticulocytes | 0.13 (0.211)

45. Secondary Outcome: Absolute Values of Reticulocytes
Description: Blood samples were collected at indicated timepoints for analysis of hematology parameter like reticulocytes. Baseline was defined as Day -1.
Time Frame: Baseline (Day -1) and Day 3
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Percentage of reticulocytes
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Percentage of reticulocytes
  Baseline (Day -1) | 1.47 (0.460)
  Day 3 | 1.59 (0.491)

46. Secondary Outcome: Change From Baseline in Blood Urea Nitrogen (BUN), Glucose, Calcium, Sodium, and Potassium Levels
Description: Blood samples were collected at indicated time-points for analysis of clinical chemistry parameters like (BUN), glucose, sodium, calcium, and potassium levels. Baseline was defined as Day -1. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1) and Day 3
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimoles per Liter
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Millimoles per Liter
  Calcium | 0.0483 (0.07315)
  Glucose | -0.1908 (0.30738)
  Potassium | 0.02 (0.288)
  Sodium | 2.8 (2.46)
  BUN | 0.2901 (0.94200)

47. Secondary Outcome: Absolute Values of BUN, Glucose, Calcium, Sodium, and Potassium Levels
Description: Blood samples were collected at indicated time-points for analysis of clinical chemistry parameters like (BUN), glucose, sodium, calcium, and potassium levels. Baseline was defined as Day -1.
Time Frame: Baseline (Day -1) and Day 3
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimoles per Liter
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Millimoles per Liter
  Calcium, Baseline (Day -1) | 2.3079 (0.08098)
  Calcium, Day 3 | 2.3562 (0.06440)
  Glucose, Baseline (Day -1) | 5.5163 (0.40684)
  Glucose, Day 3 | 5.3255 (0.39014)
  Potassium, Baseline (Day -1) | 4.18 (0.284)
  Potassium, Day 3 | 4.19 (0.124)
  Sodium, Baseline (Day -1) | 137.1 (1.88)
  Sodium, Day 3 | 139.8 (2.37)
  BUN, Baseline (Day -1) | 4.1948 (1.01395)
  BUN, Day 3 | 4.4848 (0.99251)

48. Secondary Outcome: Change From Baseline in Total and Direct Bilirubin, Creatinine and Protein Levels
Description: Blood samples were collected at indicated time-points for analysis of clinical chemistry parameters like total and direct bilirubin, creatinine and protein levels. Baseline was defined as Day -1. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1) and Day 3
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Micromoles per liter
  Total bilirubin | 3.954 (4.6188)
  Direct bilirubin | 0.428 (0.7647)
  Creatinine | 2.7072 (6.15397)
  Protein | 4.2 (3.73)

49. Secondary Outcome: Absolute Values of Total and Direct Bilirubin, Creatinine and Protein Levels
Description: Blood samples were collected at indicated time-points for analysis of clinical chemistry parameters like total and direct bilirubin, creatinine and protein levels. Baseline was defined as Day -1.
Time Frame: Baseline (Day -1) and Day 3
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Micromoles per liter
  Total bilirubin, Baseline (Day -1) | 11.008 (4.3694)
  Total bilirubin, Day 3 | 14.963 (5.2054)
  Direct bilirubin, Baseline (Day -1) | 2.565 (1.2488)
  Direct bilirubin, Day 3 | 2.993 (1.1682)
  Creatinine, Baseline (Day -1) | 80.3335 (13.88330)
  Creatinine, Day 3 | 83.0408 (13.20870)
  Protein, Baseline (Day -1) | 66.6 (3.63)
  Protein, Day 3 | 70.8 (4.57)

50. Secondary Outcome: Change From Baseline in Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) and Alkaline Phosphatase (ALP) Levels
Description: Blood samples were collected at indicated time-points for analysis of clinical chemistry parameters like AST, ALT and ALP levels. Baseline was defined as Day -1. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1) and Day 3
Population: Safety Population
Measure: Mean (Standard Deviation); unit: International units per Liter
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
International units per Liter
  ALT | 3.2 (7.46)
  AST | 0.6 (3.42)
  ALP | 0.9 (2.87)

51. Secondary Outcome: Absolute Values of AST, ALT and ALP Levels
Description: Blood samples were collected at indicated time-points for analysis of clinical chemistry parameters like AST, ALT and ALP levels. Baseline was defined as Day -1.
Time Frame: Baseline (Day -1) and Day 3
Population: Safety Population
Measure: Mean (Standard Deviation); unit: International units per Liter
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
International units per Liter
  ALT, Baseline (Day -1) | 19.4 (7.20)
  ALT, Day 3 | 22.6 (11.51)
  AST, Baseline (Day -1) | 17.9 (3.72)
  AST, Day 3 | 18.5 (4.41)
  ALP, Baseline (Day -1) | 52.3 (11.57)
  ALP, Day 3 | 53.1 (11.24)

52. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP were assessed in the supine position with a completely automated device. Day 1 (Pre-dose) was defined as Baseline. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 12
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Millimeters of mercury
  SBP | 6.2 (9.35)
  DBP | 1.6 (9.61)

53. Secondary Outcome: Absolute Values of SBP and DBP
Description: SBP and DBP were assessed in the supine position with a completely automated device. Day 1 (Pre-dose) was defined as Baseline.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 12
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Millimeters of mercury
  SBP, Day 1, Pre-dose | 107.0 (7.43)
  SBP, Day 12 | 113.2 (10.89)
  DBP, Day 1, Pre-dose | 70.1 (7.58)
  DBP, Day 12 | 71.7 (11.29)

54. Secondary Outcome: Change From Baseline in Pulse Rate
Description: Pulse rate was assessed in the supine position with a completely automated device. Day 1 (Pre-dose) was defined as Baseline. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 12
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Beats per minute | 8.7 (10.32)

55. Secondary Outcome: Absolute Values of Pulse Rate
Description: Pulse rate was assessed in the supine position with a completely automated device. Day 1 (Pre-dose) was defined as Baseline.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 12
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Beats per minute
  Day 1, Pre-dose | 58.0 (9.87)
  Day 12 | 66.7 (10.00)

56. Secondary Outcome: Change From Baseline in Body Temperature
Description: Body temperature were assessed at indicated time-points. Day 1 (Pre-dose) was defined as Baseline. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 12
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Degree Celsius | 0.06 (0.453)

57. Secondary Outcome: Absolute Values of Body Temperature
Description: Body temperature were assessed at indicated time-points. Day 1 (Pre-dose) was defined as Baseline.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 12
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | DTG/RPV 50mg/25mg FDC
Number analyzed (Participants) | 16
Degree Celsius
  Day 1, Pre-dose | 36.16 (0.271)
  Day 12 | 36.21 (0.443)

ADVERSE EVENTS:
Time Frame: Non-serious AEs and SAEs were collected from the start of the study treatment up to Day 18
Description: Non-serious AEs and SAEs were reported for the safety population which comprised of all participants who were enrolled in the study and received at least one dose of study drug.
Arm/Group | DTG/RPV 50mg/25mg FDC
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 2/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DTG/RPV 50mg/25mg FDC (N=16)
Vomiting (Gastrointestinal disorders) | 1
Vessel puncture site bruise (General disorders) | 1
Headache (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-04-04): https://cdn.clinicaltrials.gov/large-docs/38/NCT03984838/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-13): https://cdn.clinicaltrials.gov/large-docs/38/NCT03984838/SAP_001.pdf